CLINICAL TRIAL: NCT06211868
Title: Redirecting Immune, Lipid and Metabolic Drivers of Early Cardiovascular Disease: The RESET Cohort Study
Acronym: RESET
Status: Recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: RESET
Record Dates: First submitted 2023-12-06; First posted 2024-01-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational cohort
- Randomised cohort
  Interventions: Behavioral: Digital wearable and AI-human symbiotic lifestyle intervention

INTERVENTIONS:
Behavioral: Digital wearable and AI-human symbiotic lifestyle intervention — Digital wearable and AI-human symbiotic lifestyle intervention
  Groups: Randomised cohort

SUMMARY:
Project RESET is a Singapore National Medical Research Council Large Collaborative Grant funded program that brings together a nationwide community of cardiovascular, metabolic, and digital health researchers, as well as clinicians across primary and tertiary care to study the immune, lipid and metabolic drivers of early cardiovascular disease. RESET incorporates a nested randomised controlled trials (RCT) to test the use of a combined digital wearable and AI-human symbiotic lifestyle intervention to halt or reverse the progression of early disease.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 years old
* ASCVD (atherosclerotic cardiovascular disease) score of 5% and higher

Exclusion Criteria:

* Previous major cardiovascular disease (myocardial infarction, heart failure, ischemic stroke)
* Limited life expectancy
* Other ongoing unstable medical conditions
* Pregnant women

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: South-East Asian population aged 40-70 years with no prior manifest atherosclerotic cardiovascular disease (ACSVD).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event | 5 years
  Composite of cardiac death, non-fatal myocardial infarction, resuscitated cardiac arrest, non-fatal ischemic stroke, congestive heart failure, coronary revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- NUS, Singapore, Singapore